CLINICAL TRIAL: NCT04464655
Title: A 10-Minute Cardiovascular Magnetic Resonance Protocol for Cardiac Disease
Status: Recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Matthias Friedrich, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2020-6128
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease; Myocarditis; Infiltrative Cardiomyopathy; Dilated Cardiomyopathy; Hypertrophic Cardiomyopathy; Aortic Valve Stenosis; Aortic Valve Regurgitation; Pericardial Effusion; Congenital Heart Disease; Vascular Anomaly
MeSH Terms: conditions — Coronary Artery Disease; Myocarditis; Cardiomyopathy, Dilated; Cardiomyopathy, Hypertrophic; Aortic Valve Stenosis; Aortic Valve Insufficiency; Pericardial Effusion; Heart Defects, Congenital; Vascular Malformations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Age: >18 y, No known current or pre-existing medical conditions that would affect the cardiovascular or respiratory system.
- Patients: Age: > 18y, Clinically indicated CMR exam

SUMMARY:
This study aims to identify and assess new CMR techniques that can improve current CMR protocols.

DETAILED DESCRIPTION:
The aim of this study is to develop a comprehensive 10-minute protocol based on function and myocardial tissue characterization without the need for contrast injection, which can be standardized for 70% of cardiac patients.

To test this 10-minute CMR protocol for its ability to significantly improve diagnostic decision-making and to reduce cost.

To test its clinical feasibility, performance and cost-effectiveness in different populations including: Non-ischemic cardiomyopathies (-)OS-CMR and Ischemic Heart Disease and CAD (+)OS-CMR

ELIGIBILITY:
Healthy Volunteers

Inclusion Criteria:

* Age: > 18y, Informed consent No known current or pre-existing significant medical conditions that would affect the cardiovascular or respiratory system

Exclusion Criteria:

* General MRI contraindications: MR- incompatible devices such as pacemakers, defibrillators, or implanted material or foreign bodies. Consumption of caffeinated drinks or foods (including cocoa and chocolate) during the 12 hours prior to the exam.Regular nicotine consumption during the last 6 months

Patients

Inclusion Criteria:

* Age: >18 y, Informed consent, Clinically indicated CMR exam

Exclusion Criteria:

* General MRI contraindications: MR- incompatible devices such as pacemakers, defibrillators, or implanted material or foreign bodies Vasoactive medication (e.g. nitro) during the 12 hours prior to the exam. Consumption of caffeinated drinks or foods (including cocoa and chocolate) during the 12 hours prior to the exam.

Regular nicotine consumption during the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of patients with suspected cardiovascular disease who are scheduled for a clinical CMR scan as part of a routine clinical work-up.
  Patients will be stratified according to the clinical indication for CMR and their suspected or known clinical diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 2130 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Primary diagnosis comparison between SMART CMR and standard CMR | 2019-2025
  (All patients) Agreement of the suggested primary diagnosis derived from SMART CMR, compared with the diagnosis established from standard CMR protocols, using the final clinical diagnosis as established by the treating physician, as a standard of truth. If the latter is not available, the conclusions based on the results of the standard CMR protocol will be used as the standard of truth.
Main finding comparison between SMART CMR and standard CMR in patients with suspected coronary artery disease | 2019-2025
  (Patients with suspected coronary artery disease:) Agreement of the main finding regarding the presence of a coronary territory at risk for inducible myocardial ischemia myocardial derived from OS-CMR, compared with standard first-pass perfusion CMR, using the coronary angiography report as a standard of truth. If the latter is not available, the conclusions based on the results of the standard CMR first pass perfusion scan will be used as the standard of truth.

SECONDARY OUTCOMES:
SMART CMR scan completion percentage | 2019-2025
  Proportion of SMART CMR scans that could be completed according to the protocol
OS-CMR scan completion percentage | 2019-2025
  Proportion of OS-CMR scans that could be completed according to the protocol
Adverse event monitoring during SMART CMR sequences | 2019-2025
  Number and proportion of reported adverse events effects during SMART CMR
Adverse event monitoring during OS-CMR sequence | 2019-2025
  Number and proportion of reported adverse events during OS-CMR
SMART CMR sequence times vs standard protocol sequence times | 2019-2025
  Observed scan time for SMART CMR compared with the standard CMR protocol
OS-CMR sequence times vs standard protocol sequence times | 2019-2025
  Observed scan time for for OS-CMR during breathing maneuvers compared with the standard CMR first-pass perfusion protocol
Cost comparison of SMART CMR vs standard CMR protocol | 2019-2025
  Total estimated cost of SMART CMR compared with the standard CMR protocol
Cost comparison of OS-CMR vs standard CMR protocol | 2019-2025
  Total cost of OS-CMR with breathing maneuvers (based on scan time) vs the standard CMR first-pass perfusion protocol (calculated from the scan time plus any other material such as contrast agents or pharmacological vasodilators)
Septal myocardial T1 vs standard myocardial T1 | 2019-2025
  Septal myocardial T1 as estimated from SMART CMR, compared with results from standard myocardial mapping
Septal myocardial T2 vs standard myocardial T2 | 2019-2025
  Septal myocardial T2 as estimated from SMART CMR, compared with results from standard myocardial mapping
Quantitative parameter comparison between SMART CMR and CINE images | 2019-2025
  Quantitative parameters relevant to the diagnosis (see Appendix: CanSCMR Recommendations for reporting CMR) measured in SMART CMR images, compared with results from standard CMR cine images
Strain measurements vs standard cine image measurements | 2019-2025
  Longitudinal and circumferential strain measurements measured in SMART CMR images, compared with results from standard CMR cine images
SMART-CMR post-stenotic peak flow vs standard CMR flow images | 2019-2025
  Post-stenotic peak flow velocity in patients with suspected valvular disease measured in SMART CMR images, compared with results from standard CMR flow images
Intra- and inter-reader reproducibility | 2019-2025
  Correlation coefficients will be obtained to evaluate the intra- and inter-reader reproducibility of all quantitative markers.
Inter- and intra-scanner variability | 2019-2025
  Inter- and intra- scanner variability as assessed by ICC and kappa

CONTACTS AND LOCATIONS:
Overall Officials: Matthias G Friedrich, MD, Principal Investigator — Research Institute of the McGill University Health Center
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada